CLINICAL TRIAL: NCT00316511
Title: A Phase 1 Multi-Center, Dose Escalation and Pharmacokinetic Study of L-NDDP (Aroplatin) in Patients With Advanced Solid Malignancies or B-Cell Lymphoma
Brief Title: Study of L-NDDP (Aroplatin) in Patients With Advanced Solid Malignancies or B-Cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Agenus Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-726-05
Record Dates: First submitted 2006-04-19; First posted 2006-04-21 (Estimated); Last update posted 2008-10-27 (Estimated); Status verified 2008-10

CONDITIONS: Malignancies; B-Cell Lymphoma
Keywords: advanced solid malignancies; B-cell lymphoma; Aroplatin; L-NDDP; MTD; advanced solid malignancies or B-cell lymphoma
MeSH Terms: conditions — Neoplasms; Lymphoma, B-Cell | interventions — bis-neodecanoato-1,2-diaminocyclohexaneplatinum(II)

INTERVENTIONS:
Drug: Aroplatin

SUMMARY:
This is a dose escalation study. Patients will be enrolled in cohorts of three patients each, and escalation of dose to the next cohort will be determined based on dose-limiting toxicity (DLT) in the previous cohort. This study aims to identify the maximum tolerated dose (MTD) of intravenous L-NDDP. Once the MTD has been determined, an additional four patients will be enrolled at that dose level. While the MTD is determined based on safety data from each cohort's first cycle of L-NDDP therapy only, patients may continue treatment with additional cycles of L-NDDP at the same dose as their starting dose until documented progression, unacceptable toxicity, or another off study criterion is met. Patients who have not met any of the off study criteria and continue to receive L-NDDP therapy at the time when MTD is determined may be allowed to change L-NDDP dose to the MTD dose level. The study will also determine the pharmacokinetic profile of L-NDDP administration. Clinical activity of L-NDDP in solid tumor patients will be assessed as tumor response using the Response Evaluation Criteria in Solid Tumors (RECIST) criteria. Clinical activity of L-NDDP in B-cell lymphoma patients will be assessed using the International Working Group recommendations.

DETAILED DESCRIPTION:
This is a dose escalation study that utilizes a constant incremental dose increase of 50 mg/m2 per cohort. Patients will be enrolled in cohorts of three patients each, and escalation of dose to the next cohort will be determined based on dose-limiting toxicity (DLT) in the previous cohort. DLT is defined as any adverse event (AE) of severity grade 3, 4 or 5 (including serious or life-threatening) considered possibly, probably or definitely related to L-NDDP (CTCAE v3.0), which occurs during cycle 1, excluding those events that occur and are completely resolved within 4-6 hours of the first dose of L-NDDP (infusion-related reactions). This study also aims to identify the maximum tolerated dose (MTD) of intravenous L-NDDP, defined as the dose level at which no more than one out of six patients has any DLT. Once the MTD has been determined, an additional four patients will be enrolled at that dose level (for a total of 10 patients at the MTD dose level). While the MTD is determined based on safety data from each cohort's first cycle of L-NDDP therapy only, patients may continue treatment with additional cycles of L-NDDP at the same dose as their starting dose until documented progression, unacceptable toxicity or another off study criterion is met. Patients who have not met any of the off study criteria and continue to receive L-NDDP therapy at the time when MTD is determined may be allowed to change L-NDDP dose to the MTD dose level. The study will also determine the pharmacokinetic profile of L-NDDP administration through whole blood, plasma, and urine samples drawn before, during, and after L-NDDP administration. Clinical activity of L-NDDP in solid tumor patients will be assessed as tumor response using the RECIST criteria. Clinical activity of L-NDDP in B-Cell lymphoma patients will be assessed using the International Working Group Recommendations.

ELIGIBILITY:
Inclusion Criteria:

1. Advanced solid malignancies or B-cell lymphoma
2. Less than or equal to 5 anti-cancer treatment regimens, which must be concluded at least four weeks prior to the first planned L-NDDP administration
3. Measurable disease
4. Eastern Cooperative Oncology Group (ECOG) performance score of 0 or 1
5. New York Heart Association (NYHA) Class I or II
6. Greater than or equal to 18 years of age
7. Absolute neutrophil count greater than or equal to 1.5 x 10^9/L
8. Platelets greater than or equal to 100 x 10^9/L
9. Creatinine less than or equal to 1.5 x upper limit of normal (ULN)
10. ALT less than 3 x ULN in absence of liver metastases; less than 5 x ULN in presence of liver metastases.
11. Hemoglobin greater than or equal to 10 g/dL
12. Total bilirubin less than or equal to 2 x ULN
13. Female of childbearing potential must have a negative serum pregnancy test
14. Male or female patients of child producing potential must agree to use contraception or avoidance of pregnancy measures during the study and for one month after the last L-NDDP dose.
15. Signed written informed consent must be obtained and documented according to ICH-GCP, the local regulatory requirements, and the rules followed at each institution.

Exclusion Criteria:

1. Known active or untreated brain metastases
2. Other ongoing systemic cancer therapies
3. Hypersensitivity to platinum compounds
4. Other active malignancies with the exception of adequately treated in-situ carcinoma of the uterine cervix, or non-melanoma skin cancer
5. A marked baseline prolongation of QT/QTc interval (e.g. repeated demonstration [at least two assessments at a minimum of 48 hours apart] of a QTc interval of > 450 for males and > 470 for females) or history of additional risk factors for torsades des pointes or use of concomitant medication prolonging the QT/QTc interval
6. Serious illness which, in the opinion of the Principal Investigator, would prevent study completion
7. Investigational therapy currently or within four weeks prior to planned first dose of L-NDDP
8. Women who are pregnant or breastfeeding will be excluded from participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2006-03; Primary Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose and dose-limiting toxicity of L-NDDP
Assess safety of L-NDDP
Determine the pharmacokinetic profile of L-NDDP

SECONDARY OUTCOMES:
Assess clinical activity

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Boston, Massachusetts
  - Houston, Texas